CLINICAL TRIAL: NCT04309305
Title: Functional and Neurophysiological Effects of a Progressive Robot Assisted Gait Intervention Early Post Stroke
Brief Title: Robotic Exoskeleton Assisted Gait Post Stroke
Acronym: RE-Assist
Status: Enrolling by invitation | Phase: Phase 1 | Type: Interventional
Sponsor: Kessler Foundation (Other)
Responsible Party: Principal Investigator, Karen J. Nolan, PhD, Co-Principal Investigator, Kessler Foundation
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R-1073-19
Record Dates: First submitted 2020-02-10; First posted 2020-03-16 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-04

CONDITIONS: CVA; Gait, Hemiplegic
MeSH Terms: conditions — Gait Disorders, Neurologic | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (3):
- Stroke RE (Experimental): After discharge from the acute rehabilitation facility, participants in the stroke RE group will participate 3 days a week for 10 weeks in robotic exoskeleton gait training provided by a trained, licensed physical therapist. Participants will be permitted to participate in additional prescribed standard physical therapy on their own.
  Interventions: Device: EksoGT™, Ekso Bionics, Berkley, CA, USA
- Stroke SOC (Active Comparator): After discharge from the acute rehabilitation facility, participants in the stroke SOC group will participate 3 days a week for 10 weeks in standard of care gait training provided by a licensed physical therapist. Participants will be permitted to participate in additional prescribed standard physical therapy on their own.
  Interventions: Other: Standard of Care
- Healthy Control (Other): Participants in the healthy control group will not participate in any gait training. Healthy control participants will only be asked to complete 3 testing sessions.
  Interventions: Other: No Intervention

INTERVENTIONS:
Device: EksoGT™, Ekso Bionics, Berkley, CA, USA — The Robotic Exoskeleton is a device that will be strapped to the chest and legs and worn over the shoulders like a backpack that will assist in walking.
  Arms: Stroke RE
Other: Standard of Care — Standard gait therapy provided by licensed physical therapists post stroke.
  Arms: Stroke SOC
Other: No Intervention — Testing Only
  Arms: Healthy Control

SUMMARY:
The current investigation takes advantage of both a progressive and adaptive assist-as-needed massed practice and time-sensitive neuroplasticity through exoskeleton assisted walking in order to induce greater recovery-oriented CNS plasticity and consequent gains in more independent walking.

DETAILED DESCRIPTION:
The purpose of this research study is to assess whether using a wearable device, called the robotic exoskeleton (RE), can be helpful in improving recovery of walking in adults who have recently had a stroke. The study will compare the walking abilities of people who went through standard of care treatment after a stroke to those who used the robotic exoskeleton as part of their rehabilitation. This study will also look at the effects walking in the RE has on brain activity. The name of the robotic exoskeleton that is being used in this study is the EksoTM.

ELIGIBILITY:
Inclusion Criteria:

* Stroke survivors < 4 weeks from most recent stroke.
* Age: 21- 80 years
* Unilateral hemiparesis
* Medical clearance by the Medical Director
* Be able to physically fit into the exoskeleton device.
* Have joint range of motion within normal functional limits for ambulation.
* Have sufficient strength to use the hemiwalker, cane or walker (etc. assistive device) while wearing the RE.
* Patient cognitive status and ability to communicate in English must be at a level consistent with that required to participate in standard motor rehabilitation, e.g. can follow directions.
* Adequate cognitive function to give informed consent, understand the training, instructions, use investigational devices and give adequate feedback.
* No history of injury or pathology to the unaffected limb.
* physically fit within the RE: Height below 60" or above 76" and weight above 220 lbs.

Exclusion Criteria:

* Any medical issue that precludes full weight bearing and ambulation (e.g. orthopedic injuries, pain, severe spasticity).
* Skin issues that would prevent wearing the device.
* Pre-existing condition that caused exercise intolerance.(Documented uncontrolled hypertension, coronary artery disease, cardiac arrhythmia, or congestive heart failure)
* Hospitalization for heart attack, heart surgery or acute heart failure within 3 months of enrollment in study.
* Severe cognitive or psychiatric problems as well as incontinence might be contraindications to start training with a RE.
* History of severe cardiac disease such as myocardial infarction, congestive heart failure
* Uncontrolled seizure disorder.
* Uncontrolled spasticity or joint contracture that would interfere with walking in the RE and limits normal ROM during ambulation with assistive devices.
* Neuromuscular or neurological pathologies (e.g., Parkinson's disease, spinal cord injury, or traumatic brain injury with evidence of motor weakness and multiple sclerosis) that will interfere with neuromuscular function, ambulation, or limit the range of motion of the lower limbs
* Orthopedic pathologies or history that will interfere with ambulation or limit the ROM of the lower limbs (e.g., knee replacement, fixed contractures, inflammation)
* Any metal implants that are NOT MRI-compatible

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2020-01-30 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Functional Independence Measure (FIM) (aim 1) | Change from Baseline FIM at 10 weeks
  a conventional assessment measure of motor function
Within-brain functional connectivity (aim 2) | Change from Baseline Within-brain functional connectivity at 10 weeks
  fMRI connectivity between selected regions of interest within the sensorimotor and attention networks.
TMS recruitment curve slope (aim 3) | Change from Baseline TMS recruitment curve slope at 10 weeks
  A recruitment curve created using measure of primary motor cortex Motor Evoked Potential (MEP) at several stimulation thresholds.
electroencephalogram (EEG) (aim 3) | Change from Baseline EEG at 10 weeks
  a measure of brain activation at different phases of gait cycle (swing versus double support).
electromyography (EMG) (aim 3) | Change from Baseline EMG at 10 weeks
  a measure of muscle activation (EMG signal) at different phases of gait cycle (swing versus double support).
10MWT (aims 1-3) | Change from Baseline 10MWT at 10 weeks
  10 meters walking test to evaluate walking speedafter stroke and in response to the intervention.
6MWT (aims 1-3) | Change from Baseline 6MWT at 10 weeks
  6 minutes walking test to evaluate endurancein connectivity after stroke and in response to the intervention.
TUG (aims 1-3) | Change from Baseline TUG at 10 weeks
  time up and go (TUG) test
structural connectivity (aim 2) | Change from Baseline structural connectivity at 10 weeks
  Diffusion Tensor Imaging (DTI) and fractal dimensions (FD) measures of structural connectivity

CONTACTS AND LOCATIONS:
Overall Officials: Karen J. Nolan, PhD, Principal Investigator — Kessler Foundation; Soha Saleh, PhD, Principal Investigator — Kessler Foundation
Locations (1):
- Kessler Foundation, West Orange, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No